CLINICAL TRIAL: NCT00393354
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week Trial to Assess the Efficacy and Safety of MK0663 in Patients With Chronic Low Back Pain
Brief Title: Effect of Etoricoxib to Treat Chronic Low Back Pain (0663-041)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-041; 2006_548
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, Etoricoxib / Duration of Treatment : 12 Weeks
Drug: Comparator : placebo (unspecified) /Duration of Treatment : 12 Weeks

SUMMARY:
Study the effect of etoricoxib 60 mg and 90 mg compared to placebo to treat chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for previous 3 months and majority of days in last month
* Regular use of acetaminophen or NSAID to treat low back pain in past month
* Judged to be in otherwise good health

Exclusion Criteria:

* Low back pain that is due to secondary causes
* Radicular/myelopathic pain
* Surgery for low back pain within the past 6 months
* Active lawsuit or claim pertaining to their low back pain
* Disease that may confound the results of the study or pose risk to the patients
* Corticosteroid use in past month
* Previous participation in MK0663 study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2000-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Low back pain intensity scale (0-100 mm VAS) over 4 weeks compared to placebo

SECONDARY OUTCOMES:
Low back pain intensity scale (0-100 mm VAS) over 12 weeks compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Pallay RM, Seger W, Adler JL, Ettlinger RE, Quaidoo EA, Lipetz R, O'Brien K, Mucciola L, Skalky CS, Petruschke RA, Bohidar NR, Geba GP. Etoricoxib reduced pain and disability and improved quality of life in patients with chronic low back pain: a 3 month, randomized, controlled trial. Scand J Rheumatol. 2004;33(4):257-66. doi: 10.1080/03009740410005728. PMID 15370723
- [Background] Curtis SP, Ng J, Yu Q, Shingo S, Bergman G, McCormick CL, Reicin AS. Renal effects of etoricoxib and comparator nonsteroidal anti-inflammatory drugs in controlled clinical trials. Clin Ther. 2004 Jan;26(1):70-83. doi: 10.1016/s0149-2918(04)90007-0. PMID 14996519
- [Background] Sheldon EA, Bird SR, Smugar SS, Tershakovec AM. Correlation of measures of pain, function, and overall response: results pooled from two identical studies of etoricoxib in chronic low back pain. Spine (Phila Pa 1976). 2008 Mar 1;33(5):533-8. doi: 10.1097/BRS.0b013e3181657d24. PMID 18317199